CLINICAL TRIAL: NCT02272790
Title: A Multicentre Phase II Study of Adavosertib Plus Chemotherapy in Patients With Platinum-Resistant Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Adavosertib Plus Chemotherapy in Platinum-Resistant Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6010C00004; GYN 49 (Other: Sarah Cannon Development Innovations); 2015-000886-30 (EudraCT Number)
Record Dates: First submitted 2014-10-14; First posted 2014-10-23 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-08

CONDITIONS: Ovarian, Fallopian Tube, Peritoneal Cancer, P53 Mutation
Keywords: Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
MeSH Terms: interventions — adavosertib; Paclitaxel; Carboplatin; Gemcitabine; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (adavosertib + gemcitabine) (Experimental): Adavosertib (175 mg PO) will be taken on Days 1-2, 8-9, and 15-16. Gemcitabine 800 mg/m² will be administered IV on days 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: Adavosertib; Drug: Gemcitabine
- Arm B (adavosertib + paclitaxel) (Experimental): Five doses of adavosertib (225 mg PO BID) will be taken in approximate 12 hour intervals over 2.5 days weekly (Days 1-3, 8-10, and 15-17). Weekly paclitaxel 80 mg/m² IV will be administered according to institutional standards on Day 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: Adavosertib; Drug: Paclitaxel
- Arm C/C2 (adavosertib + carboplatin) (Experimental): Arm C: Five doses of adavosertib (225 mg PO BID) will be taken in approximate 12 hour intervals over 2.5 days (Days 1-3). Carboplatin AUC 5 IV will be administered according to institutional standards on Day 1 of each 21-Day cycle.
  Arm C2: Five doses of adavosertib (225 mg PO BID) 2.5 days per dosing week (QW), on Weeks 1 (D1-3), 2 (D8-10) and 3 (D15-17), or on Weeks 1 (D1-3) and 2 (D8-10) ( 2 weeks on followed by 1 week off.) Carboplatin AUC 5 IV will be administered according to institutional standards on Day 1 of each 21 day cycle.
  Interventions: Drug: Adavosertib; Drug: Carboplatin
- Arm D (adavosertib + PLD) (Experimental): Five doses of adavosertib (175 mg or 225 mg) will be taken in approximate 12 hour intervals over 2.5 days (Days 1, 2, and 3) of each 28-day cycle. PLD will administered IV on Day 1 of each cycle.
  Interventions: Drug: Adavosertib; Drug: PLD

INTERVENTIONS:
Drug: Adavosertib — Adavosertib will be taken as oral capsules with water, approx. 2 hours before or 2 hours after food.
  Other Names: MK1775
Drug: Paclitaxel — Paclitaxel will be administered as a 1-hour IV infusion (± 10 minutes) at a dose of 80 mg/m2 according to institutional standards on Days 1, 8, and 15 of each 28 Day cycle.
  Patients should be pre-medicated with corticosteroids, diphenhydramine and/or H2 antagonists according to institutional standards.
  Other Names: Taxol
  Arms: Arm B (adavosertib + paclitaxel)
Drug: Carboplatin — Carboplatin, at a dose calculated to produce an AUC of 5 will be administered by intravenous infusion according to institutional standards on Day 1 of each 21 Day cycle. The carboplatin dose will be calculated using the Calvert Formula based on the patient's glomerular filtration rate (GFR) which is estimated by using the creatinine clearance.
  Other Names: Paraplatin
  Arms: Arm C/C2 (adavosertib + carboplatin)
Drug: Gemcitabine — Gemcitabine 800 mg/m² will be administered IV on Days 1, 8, and 15 of each 28-Day cycle.
  Arms: Arm A (adavosertib + gemcitabine)
Drug: PLD — PLD (pegylated liposomal doxorubicin) 40 mg/m² IV will be given on Day 1 of each 28-Day cycle.
  Arms: Arm D (adavosertib + PLD)

SUMMARY:
Adavosertib in combination with carboplatin, paclitaxel, gemcitabine, or PLD.

DETAILED DESCRIPTION:
This is an open-label, four-arm lead-in safety and efficacy study in which adavosertib will be combined in four separate treatment arms as follows: adavosertib plus gemcitabine (Arm A); adavosertib plus weekly paclitaxel (Arm B); adavosertib plus carboplatin (Arm C); and adavosertib plus PLD (Arm D). A subset of patients will be evaluated for the safety assessment of each treatment arm.

The adavosertib plus paclitaxel arm (Arm B) will enrol approximately 30 additional patients at selected sites as part of a further efficacy evaluation based on emerging data that suggests clinical activity.

In addition, the adavosertib plus carboplatin arm (Arm C) will enrol approximately 23 patients overall at selected sites as part of a further efficacy evaluation based on emerging data that suggests clinical activity.

To further optimise the dosing schedule of adavosertib in Arm C, a safety expansion arm (referred to as Arm C2) of approximately 12 additional patients will be enrolled at selected sites to explore emerging pre-clinical and clinical data that suggest that prolonged adavosertib exposure may increase the clinical activity.

ELIGIBILITY:
Inclusion

* Has read and understands the informed consent form (ICF) and has given written IC prior to any study specific procedures.
* Histologic or cytologic diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Progressed within 6 months of completing at least 4 cycles of a first-line platinum-containing regimen for Stage III/IV disease. Patients with refractory disease (progression during platinum-containing therapy) are ineligible.
* No more than 2-4 prior treatment regimens for Stage III/IV disease, defined as investigational, chemotherapy, hormonal, biologic, or targeted therapy.
* Prior doxorubicin (or other anthracycline) at a cumulative dose of ≤ 360 mg/m² or cumulative epirubicin dose of ≤ 720 mg/m² (calculated using doxorubicin equivalent doses: 1 mg of doxorubicin = 1 mg PLD = 0.3 mg mitoxantrone = 0.25 mg idarubicin). Subjects without any prior anthracycline exposure can also be included. Applies to Arm D only.
* At least 1 measurable lesion according to RECIST v1.1.
* Any prior palliative radiation therapy must be completed at least 7 days prior to start of study treatment and patients must have recovered from any acute adverse effects prior to start of study treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 - 1.
* Baseline Laboratory Values:

  1. ANC ≥1500/μL
  2. HgB ≥ 9 g/dL with no blood transfusions in the past 28 days
  3. Platelets ≥ 100,000/μL
  4. ALT & AST ≤3 x ULN or ≤5 x ULN if known hepatic metastases
  5. Serum bilirubin within normal limits (WNL) or ≤1.5 x the ULN in patients with liver metastases; or total bilirubin ≤3.0 x ULN with direct bilirubin WNL in patients with well documented Gilbert's Syndrome.
  6. Serum creatinine ≤1.5 x the ULN and a calculated creatinine clearance (CrCl) ≥45 mL/min by the Cockcroft-Gault method.
* Left ventricular ejection fraction (LVEF) WNL of the institution as determined by multiple uptake gated acquisition (MUGA) or echocardiography (ECHO) (applies to Arm D only).
* Female patients, ≥18, (not of childbearing potential and fertile female patients of childbearing potential) who agree to use adequate contraceptive measures from 2 weeks prior to the study and until 1 month after study treatment discontinuation, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to start.
* Predicted life expectancy ≥ 12 weeks

Exclusion

* Use of a study drug (approved or investigational drug therapy) ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of study treatment. For study drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the study drug and administration of study treatment is required.
* Major surgical procedures ≤ 28 days of beginning study, or minor surgical procedures ≤ 7 days. No waiting period following port-a-cath placement, or any other central venous access placement.
* Grade >1 toxicity from prior therapy (except alopecia or anorexia).
* Known malignant CNS disease other than neurologically stable, treated brain metastases, defined as metastasis having no evidence of progression or haemorrhage after treatment for at least 2 weeks (including brain radiotherapy). Must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrolment.
* Patient has had prescription or non-prescription drugs or other products (i.e. grapefruit juice) known to be sensitive CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors or inducers of CYP3A4 which cannot be discontinued 2 weeks prior to Day 1 of dosing and withheld throughout the study until 2 weeks after last dose of study drug.
* Caution should be exercised when inhibitors or substrates of P-gP, substrates of CYP1A2 with a narrow therapeutic range, sensitive substrates of CYP2C19 or CYP2C19 substrates with a narrow therapeutic range are administered with adavosertib.
* Herbal medications should be discontinued 7 days prior to the first dose of study treatment.
* Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) ≥ Class 2:

  1. Unstable angina pectoris
  2. Congestive heart failure
  3. Acute myocardial infarction
  4. Conduction abnormality not controlled with pacemaker or medication
  5. Significant ventricular or supraventricular arrhythmias (patients with chronic rate controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
* Adavosertib should not be given to patients who have a history of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected. Adavosertib has not been studied in patients with ventricular arrhythmias or recent myocardial infarction.
* Corrected QT interval (QTc) >470 msec at study entry or congenital long QT syndrome.
* Pregnant or lactating.
* Serious active infection at the time of enrolment, or another serious underlying medical condition that would impair the patient's ability to receive study treatment.
* Presence of other active cancers, or history of treatment for invasive cancer within 3 years. Patients with Stage I cancer who have received definitive local treatment within 3 years, and whom are considered unlikely to recur, are eligible. Patients with previously treated in-situ carcinoma (i.e., non-invasive) are eligible, as are patients with prior non-melanoma skin cancers.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, MD, Principal Investigator — Stephenson Cancer Center, University of Oklahoma Health Sciences Center
Locations (19):
- United States (17):
  - Research Site, Gilbert, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Abington, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Milwaukee, Wisconsin
- Research Site, Toronto, Ontario, Canada
- Research Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Moore KN, Chambers SK, Hamilton EP, Chen LM, Oza AM, Ghamande SA, Konecny GE, Plaxe SC, Spitz DL, Geenen JJJ, Troso-Sandoval TA, Cragun JM, Rodrigo Imedio E, Kumar S, Mugundu GM, Lai Z, Chmielecki J, Jones SF, Spigel DR, Cadoo KA. Adavosertib with Chemotherapy in Patients with Primary Platinum-Resistant Ovarian, Fallopian Tube, or Peritoneal Cancer: An Open-Label, Four-Arm, Phase II Study. Clin Cancer Res. 2022 Jan 1;28(1):36-44. doi: 10.1158/1078-0432.CCR-21-0158. Epub 2021 Oct 13. PMID 34645648
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6010C00004&attachmentIdentifier=617d4afb-03ad-4dac-9100-8ce0250343b6&fileName=D6010C00004_Statistical_Analysis_Plan_v5.0_redact-_Final_pdfa.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6010C00004&attachmentIdentifier=ed07c4a3-8013-4481-a040-47104f414937&fileName=d6010c00004-csp-amendment-10-redact-_Final_pdfa.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6010C00004&attachmentIdentifier=6c837a44-25f7-4e56-8466-debf040a850f&fileName=d6010c00004-study-synopsis-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multi-center study was conducted at 20 sites: 18 in the USA, 1 in Canada, and 1 in The Netherlands. Ninety-five (95) patients were enrolled; 94 patients received treatment. The first patient started treatment on 2 Feb 2015; the final patients were still receiving treatment and were censored at the time of database lock on 14 Dec 2018.
Pre-assignment Details: One hundred twenty-six (126) patients consented and underwent screening; 94 patients passed screening, whereas 32 patients failed screening tests and were not eligible. The Full Analysis Set consists of 94 patients.
Groups:
- Arm A: Adavosertib 175 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of 28 day cycles.
  Gemcitabine 800 mg/m² IV on Days 1, 8, and 15 of 28 day cycles.
- Arm B: Adavosertib 225 mg orally BID (5 doses over 3 days) on Days 1-3, 8-10, and 15-17 of 28 day cycles.
  Paclitaxel 80 mg/m² IV on Days 1, 8, and 15 of 28 day cycles.
- Arm C: Adavosertib 225 mg orally BID (5 doses over 3 days) on Days 1-3 of 21 day cycles.
  Carboplatin AUC 5 IV on Day 1 of 21 day cycles.
- Arm C2: Adavosertib 225 mg orally BID (5 doses over 3 days) on Days 1-3, 8-10, and 15-17 of 21 day cycles.
  Carboplatin AUC 5 IV on Day 1 of 21 day cycles.
- Arm D-175 mg: Adavosertib 175 mg orally BID (5 doses over 3 days) on Days 1-3 of 28 day cycles.
  Pegylated liposomal doxorubicin 40 mg/m² IV on Day 1 of 28 day cycles.
- Arm D-225 mg: Adavosertib 225 mg orally BID (5 doses over 3 days) on Days 1-3 of 28 day cycles.
  Pegylated liposomal doxorubicin 40 mg/m² IV on Day 1 of 28 day cycles.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Started | 9 | 39 | 23 | 12 | 6 | 6
Completed | 9 | 38 | 23 | 12 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg | Total
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.75) | 60.9 (8.16) | 62.1 (11.29) | 60.3 (6.96) | 57.3 (14.58) | 61.0 (7.16) | 60.7 (9.30)
Age, Continuous [Median (Full Range); unit: years] | 63.0 [46 to 72] | 60.0 [45 to 76] | 62.0 [34 to 85] | 58.5 [52 to 76] | 58.5 [40 to 72] | 60.5 [54 to 70] | 60.0 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 38 | 23 | 12 | 6 | 6 | 94
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 2 | 2 | 0 | 1 | 12
  Not Hispanic or Latino | 8 | 31 | 21 | 10 | 5 | 5 | 80
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 0 | 0 | 0 | 8
  White | 7 | 24 | 20 | 10 | 6 | 6 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 1 | 2 | 0 | 0 | 8
Region of Enrollment [Number; unit: Participants]
  United States | 7 | 30 | 23 | 12 | 6 | 6 | 84
  Canada | 2 | 7 | 0 | 0 | 0 | 0 | 9
  Netherlands | 0 | 1 | 0 | 0 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  < 65 | 5 | 26 | 14 | 8 | 3 | 3 | 59
  ≥ 65 | 4 | 12 | 9 | 4 | 3 | 3 | 35
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out light or sedentary work; 2 = Ambulatory and capable of all self care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, cannot carry on any self care. Totally confined to bed or chair; 5 = Dead.
  Participants
    PS = 0 | 5 | 19 | 13 | 4 | 1 | 3 | 45
    PS = 1 | 4 | 19 | 10 | 8 | 5 | 3 | 49
    PS = 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    PS = 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    PS = 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Time from 1st positive biopsy for disease to consent for this study (mean) [Mean (Standard Deviation); unit: Weeks] | 52.0 (11.83) | 70.9 (46.42) | 62.3 (24.68) | 86.1 (55.67) | 61.4 (23.88) | 65.8 (20.82) | 68.0 (38.93)
Time from 1st positive biopsy for disease to consent for this study (median) [Median (Full Range); unit: Days] | 49.9 [35.9 to 77.1] | 54.9 [31.4 to 250.4] | 54.1 [30.0 to 113.6] | 74.9 [25.1 to 241.0] | 62.9 [30.6 to 87.4] | 71.1 [41.1 to 90.0] | 54.9 [25.1 to 250.4]
Local or Regional Recurrence [Count of Participants; unit: Participants]
  Yes | 5 | 26 | 17 | 9 | 4 | 6 | 67
  No | 4 | 12 | 6 | 3 | 2 | 0 | 27
Time from local/regional recurrence to consent for this study (mean) [Mean (Standard Deviation); unit: Weeks] — Sixty-seven (67) patients has a local or regional recurrence. Population: Sixty-seven (67) patients has a local or regional recurrence.
  Weeks
    number analyzed (Participants) | 5 | 26 | 17 | 9 | 4 | 6 | 67
    (all) | 12.2 (14.98) | 34.3 (51.20) | 20.6 (20.23) | 47.0 (57.13) | 39.3 (27.78) | 5.2 (3.61) | 28.6 (41.11)
Time from local/regional recurrence to consent for this study (median) [Median (Full Range); unit: Weeks] — Sixty-seven (67) patients has a local or regional recurrence. Population: Sixty-seven (67) patients has a local or regional recurrence.
  Weeks
    number analyzed (Participants) | 5 | 26 | 17 | 9 | 4 | 6 | 67
    (all) | 6.1 [3.0 to 38.9] | 18.6 [0.6 to 200.4] | 16.6 [1.6 to 70.6] | 15.4 [0.9 to 177.9] | 37.7 [7.6 to 74.3] | 5.6 [0.4 to 10.0] | 13.0 [0.4 to 200.4]
Distant Metastases [Count of Participants; unit: Participants]
  Yes | 3 | 29 | 11 | 12 | 5 | 5 | 65
  No | 6 | 9 | 12 | 0 | 1 | 1 | 29
Histology [Count of Participants; unit: Participants]
  Serous Epithelial Carcinoma | 9 | 33 | 21 | 12 | 4 | 6 | 85
  Endometrioid Carcinoma | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Clear Cell Epithelial Carcinoma | 0 | 2 | 1 | 0 | 1 | 0 | 4
  Transitional Cell/Brenner Carcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Squamous Cell Epithelial Carcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Undifferentiated Epithelial Carcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mucinous Epithelial Carcinoma | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Mixed Epithelial Carcinoma | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Missing | 0 | 1 | 1 | 0 | 0 | 0 | 2
Histological Grade [Count of Participants; unit: Participants]
  G1 - Well Differentiated | 1 | 1 | 0 | 2 | 0 | 0 | 4
  G2 - Moderately Differentiated | 0 | 1 | 1 | 0 | 0 | 0 | 2
  G3 - Poorly Differentiated | 5 | 28 | 15 | 9 | 5 | 3 | 65
  G4 - Undifferentiated | 0 | 3 | 2 | 0 | 1 | 1 | 7
  GX - Grade cannot be assessed or Not Applicable | 2 | 3 | 3 | 1 | 0 | 2 | 11
  Missing | 1 | 2 | 2 | 0 | 0 | 0 | 5
Stage at Initial Diagnosis [Count of Participants; unit: Participants]
  IC | 0 | 1 | 0 | 0 | 0 | 0 | 1
  IIC | 0 | 0 | 0 | 0 | 1 | 0 | 1
  III | 0 | 1 | 1 | 0 | 0 | 0 | 2
  IIIA | 0 | 1 | 0 | 0 | 1 | 0 | 2
  IIIB | 0 | 2 | 0 | 0 | 1 | 0 | 3
  IIIC | 6 | 14 | 14 | 4 | 1 | 5 | 44
  IV | 3 | 18 | 8 | 8 | 2 | 1 | 40
  Missing | 0 | 1 | 0 | 0 | 0 | 0 | 1
Metastatic Disease [Count of Participants; unit: Participants]
  Yes | 7 | 37 | 19 | 12 | 5 | 6 | 86
  No | 2 | 1 | 4 | 0 | 1 | 0 | 8
Sites of Metastatic Disease [Number; unit: Participants]
  Bone | 2 | 1 | 0 | 0 | 0 | 0 | 3
  Breast | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Distant Lymph Nodes | 1 | 14 | 10 | 8 | 3 | 1 | 37
  Liver | 6 | 13 | 4 | 3 | 2 | 3 | 31
  Local or Regional Lymph Nodes | 4 | 20 | 12 | 7 | 1 | 1 | 45
  Lung | 1 | 10 | 3 | 2 | 1 | 2 | 19
  Other | 4 | 31 | 8 | 9 | 5 | 2 | 59
  Skin or Subcutaneous | 0 | 1 | 0 | 0 | 0 | 0 | 1
Prior Systemic Therapy [Count of Participants; unit: Participants]
  Yes | 9 | 38 | 23 | 12 | 6 | 6 | 94
  No | 0 | 0 | 0 | 0 | 0 | 0 | 0
Time from end of most recent prior systemic therapy to consent for this trial (mean) [Mean (Standard Deviation); unit: Weeks] | 11.0 (9.54) | 14.4 (15.45) | 10.5 (7.81) | 15.4 (15.12) | 12.9 (11.36) | 13.4 (12.08) | 13.1 (12.75)
Time from end of most recent prior systemic therapy to consent for this trial (median) [Median (Full Range); unit: Weeks] | 5.4 [2 to 25] | 6.9 [1 to 82] | 6.9 [0 to 27] | 9.4 [2 to 53] | 10.5 [2 to 32] | 12.2 [1 to 36] | 7.6 [0 to 82]
Number of prior treatment regimens [Count of Participants; unit: Participants]
  0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 | 3 | 12 | 8 | 4 | 3 | 2 | 32
  2 | 6 | 16 | 9 | 5 | 3 | 4 | 43
  3 | 0 | 10 | 6 | 2 | 0 | 0 | 18
  >3 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Disease setting for most recent prior regimen [Count of Participants; unit: Participants]
  Neoadjuvant | 0 | 4 | 2 | 2 | 0 | 1 | 9
  Adjuvant | 4 | 15 | 13 | 4 | 4 | 1 | 41
  Metastatic | 5 | 19 | 8 | 6 | 2 | 4 | 44
Disease setting for most recent prior regimen [Count of Participants; unit: Participants]
  Adj/Neoadj in Localized disease (Stage I or II) | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Adjuvant in advanced disease (Stage III or IV) | 4 | 14 | 13 | 4 | 3 | 1 | 39
  Neoadjuvant in advanced disease (Stage III or IV) | 0 | 3 | 2 | 2 | 0 | 1 | 8
  Metastatic | 5 | 19 | 8 | 6 | 2 | 4 | 44
  Missing | 0 | 1 | 0 | 0 | 0 | 0 | 1
Best overall response to most recent prior regimen [Count of Participants; unit: Participants]
  Complete Response (CR) | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Partial Response (PR) | 0 | 2 | 1 | 1 | 0 | 1 | 5
  Non-CR/Non-PD | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Stable Disease (SD) | 2 | 4 | 1 | 2 | 1 | 0 | 10
  Progressive Disease (PD) | 2 | 9 | 5 | 4 | 1 | 2 | 23
  Not Evaluable | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Applicable | 5 | 21 | 16 | 5 | 3 | 1 | 51
Reason most recent prior regimen ended [Count of Participants; unit: Participants]
  Completed planned treatment | 4 | 14 | 10 | 5 | 3 | 2 | 38
  Progressive Disease | 5 | 19 | 10 | 7 | 2 | 3 | 46
  Toxicity | 0 | 3 | 1 | 0 | 1 | 1 | 6
  Other | 0 | 2 | 2 | 0 | 0 | 0 | 4
Prior Surgery [Count of Participants; unit: Participants]
  Yes | 8 | 35 | 22 | 11 | 6 | 6 | 88
  No | 1 | 3 | 1 | 1 | 0 | 0 | 6
Prior Radiotherapy [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 0 | 0 | 0 | 0 | 1
  No | 9 | 37 | 23 | 12 | 6 | 6 | 93
Weight (mean) [Mean (Standard Deviation); unit: Kilograms] | 73.5 (21.56) | 73.2 (15.89) | 75.7 (19.25) | 70.6 (9.45) | 70.2 (14.11) | 65.7 (8.61) | 72.8 (16.12)
Weight (median) [Median (Full Range); unit: Kilograms] | 69.6 [47.6 to 124.1] | 69.6 [47.4 to 117.6] | 71.5 [44.8 to 114.0] | 67.7 [56.9 to 85.1] | 68.2 [56.2 to 95.1] | 67.8 [51.1 to 74.4] | 69.7 [44.8 to 124.1]
Systolic Blood Pressure (mean) [Mean (Standard Deviation); unit: mmHg] | 130.0 (15.23) | 125.2 (13.37) | 127.7 (10.65) | 122.3 (6.40) | 125.2 (17.22) | 127.5 (9.35) | 126.1 (12.16)
Systolic Blood Pressure (median) [Median (Full Range); unit: mmHg] | 130.0 [109.0 to 153.0] | 126.5 [100.0 to 159.0] | 128.0 [110.0 to 153.0] | 121.0 [115.0 to 137.0] | 120.0 [112.0 to 159.0] | 126.5 [113.0 to 142.0] | 126.0 [100.0 to 159.0]
Diastolic Blood Pressure (mean) [Mean (Standard Deviation); unit: mmHg] | 76.2 (10.96) | 76.7 (7.74) | 74.8 (8.03) | 74.4 (8.26) | 73.0 (6.66) | 78.7 (6.02) | 75.8 (7.99)
Diastolic Blood Pressure (median) [Median (Full Range); unit: mmHg] | 78.0 [62.0 to 90.0] | 78.0 [59.0 to 93.0] | 75.0 [61.0 to 95.0] | 73.5 [62.0 to 87.0] | 74.0 [63.0 to 83.0] | 77.5 [73.0 to 89.0] | 76.0 [59.0 to 95.0]
Body Surface Area (mean) [Mean (Standard Deviation); unit: m²] | 1.8 (0.25) | 1.8 (0.19) | 1.8 (0.22) | 1.8 (0.13) | 1.8 (0.18) | 1.7 (0.10) | 1.8 (0.19)
Body Surface Area (median) [Median (Full Range); unit: m²] | 1.8 [1.5 to 2.3] | 1.8 [1.4 to 2.3] | 1.8 [1.4 to 2.3] | 1.7 [1.6 to 2.0] | 1.7 [1.6 to 2.1] | 1.7 [1.5 to 1.8] | 1.7 [1.4 to 2.3]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the proportion of patients achieving a complete or partial tumour response according to RECIST v1.1 criteria.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: This analysis was conducted on the Full Analysis Set, comprised of all patients who received at least dose of study treatment (n = 94).
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 1 | 11 | 7 | 8 | 2 | 1

2. Secondary Outcome: Disease Control Rate (DCR)
Description: The Disease Control Rate is defined as the proportion of patients achieving a complete response (CR), partial response (PR), or stable disease (SD) according to RECIST v1.1 criteria.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 3 | 27 | 19 | 12 | 3 | 5

3. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) is defined as the time from first documented tumour response until the date of documented progression or death from any cause.
Time Frame: Throughout the duration of the study, approximately 19 months.
Population: Duration of Response (DoR) was calculated for all responders (N = 30)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 1 | 11 | 7 | 8 | 2 | 1
Months | 4.4 [0 to NA] — non calculable | 12.0 [3.7 to NA] — non calculable | NA [NA to NA] — non calculable | 10.4 [5.8 to NA] — non calculable | NA [NA to NA] — non calculable | NA [NA to NA] — non calculable

4. Secondary Outcome: Progression Free Survival (Median, 80% CI)
Description: Progression-free survival (PFS) was defined as the elapsed time from date of first dose of AZD1775 until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdrew from therapy or received another anti-cancer therapy prior to progression. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
  Progression-free survival was derived based on scan/assessment dates, not visit dates.
Time Frame: Throughout the Study, Approximately 4 years
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Months | 1.7 [1.6 to 5.5] | 5.5 [3.8 to 7.1] | 4.2 [3.9 to 5.6] | 12.0 [8.6 to 13.1] | 2.7 [1.7 to NA] — non calculable | NA [NA to NA] — non calculable

5. Secondary Outcome: Progression Free Survival (Median, 95% CI)
Description: as for outcome 4
Time Frame: Throughout the Study, Approximately 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Months | 1.7 [0.3 to 5.5] | 5.5 [3.7 to 7.4] | 4.2 [2.8 to 8.9] | 12.0 [2.7 to NA] — non calculable | 2.7 [0.5 to NA] — non calculable | NA [NA to NA] — non calculable

6. Secondary Outcome: Overall Survival (Median, 80% CI)
Description: Overall survival (OS) was defined as the elapsed time from the date of first dose of AZD1775 until death due to any cause. Any patient not known to have died at the time of the analysis was censored based on the last recorded date on which the patient was known to be alive.
Time Frame: Throughout the Study, Approximately 4 years
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Months | 16.0 [6.7 to NA] — non calculable | NA [15.6 to NA] — Non calculable | 8.9 [8.0 to NA] — non calculable | 19.2 [12.4 to 19.2] | 3.8 [2.0 to 6.2] | NA [NA to NA] — non calculable

7. Secondary Outcome: Overall Survival (Median, 95% CI)
Description: as for outcome 6
Time Frame: Throughout the Study, Approximately 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Months | 16.0 [2.2 to NA] — non calculable | NA [11.6 to NA] — non calculable | 8.9 [8.0 to NA] — non calculable | 19.2 [12.4 to 19.2] | 6.2 [2.0 to NA] — non calculable | NA [NA to NA] — non calculable

8. Secondary Outcome: Gynecologic Cancer Intergroup (GCIG) CA-125 Response
Description: The GCIG CA-125 response is defined as the proportion of patients achieving a 50% reduction in CA-125 levels from baseline, if baseline level is ≥2 x the upper limit of normal (ULN) within 2 weeks prior to starting treatment. Response must be confirmed and maintained for at least 28 days.
Time Frame: Throughout the study, approximately 4 years
Population: The CA-125 analysis set was comprised of all dosed patients with pre-treatment serum sample showing CA-125 ≥ 2 x ULN within 2 weeks before starting treatment.
Measure: Number (90% Confidence Interval); unit: Percent
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 8 | 28 | 15 | 11 | 4 | 4
Percent | 25.0 [4.6 to 60.0] | 53.6 [36.6 to 69.9] | 26.7 [9.7 to 51.1] | 63.6 [35.0 to 86.5] | 25.0 [1.3 to 75.1] | 25.0 [1.3 to 75.1]

9. Secondary Outcome: The Number of Patients Experiencing Treatment-emergent Adverse Events (TEAEs) by Maximum CTCAE Grade.
Description: The number of patients experiencing at least one treatment-related adverse event (TEAE) by maximum CTCAE grade.
  Severity Grade 1 = Mild; Severity Grade 2 = Moderate; Severity Grade 3 = Severe; Severity Grade 4 = Life Threatening; Severity Grade 5 = Fatal
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants
  Number of patients with ≥1 TEAE of max Grade 1 | 0 | 2 | 0 | 0 | 0 | 0
  Number of patients with ≥1 TEAE of max Grade 2 | 1 | 1 | 5 | 0 | 3 | 4
  Number of patients with ≥1 TEAE of max Grade 3 | 2 | 19 | 10 | 4 | 3 | 0
  Number of patients with ≥1 TEAE of max Grade 4 | 6 | 15 | 8 | 8 | 0 | 2
  Number of patients with ≥1 TEAE of max Grade 5 | 0 | 1 | 0 | 0 | 0 | 0

10. Secondary Outcome: The Number of Patients Experiencing Treatment-emergent Adverse Events (TEAEs) Related to Adavosertib by Maximum CTCAE Grade
Description: The number and proportion of patients experiencing at least one treatment-related adverse event (TEAE) related to adavosertib by maximum CTCAE grade
  Severity Grade 1 = Mild; Severity Grade 2 = Moderate; Severity Grade 3 = Severe; Severity Grade 4 = Life Threatening; Severity Grade 5 = Fatal
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants
  Number of patients with ≥1 TEAE of max Grade 1 | 0 | 3 | 2 | 0 | 0 | 0
  Number of patients with ≥1 TEAE of max Grade 2 | 1 | 4 | 5 | 0 | 5 | 4
  Number of patients with ≥1 TEAE of max Grade 3 | 3 | 16 | 7 | 4 | 1 | 0
  Number of patients with ≥1 TEAE of max Grade 4 | 5 | 14 | 8 | 8 | 0 | 2
  Number of patients with ≥1 TEAE of max Grade 5 | 0 | 1 | 0 | 0 | 0 | 0

11. Secondary Outcome: The Number of Patients Experiencing Treatment-emergent Adverse Events (TEAEs) Related to Chemotherapy by Maximum CTCAE Grade
Description: The number of patients experiencing at least one treatment-related adverse event (TEAE) related to chemotherapy by maximum CTCAE grade.
  Severity Grade 1 = Mild; Severity Grade 2 = Moderate; Severity Grade 3 = Severe; Severity Grade 4 = Life Threatening; Severity Grade 5 = Fatal
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants
  Number of patients with ≥1 TEAE of max Grade 1 | 0 | 4 | 0 | 0 | 0 | 0
  Number of patients with ≥1 TEAE of max Grade 2 | 1 | 5 | 6 | 0 | 5 | 4
  Number of patients with ≥1 TEAE of max Grade 3 | 3 | 13 | 8 | 4 | 1 | 0
  Number of patients with ≥1 TEAE of max Grade 4 | 5 | 15 | 8 | 8 | 0 | 2
  Number of patients with ≥1 TEAE of max Grade 5 | 0 | 1 | 0 | 0 | 0 | 0

12. Secondary Outcome: Serious Adverse Events
Description: The number of patients experiencing at least one serious adverse event (SAE).
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants
  Pts. with ≥ one serious TEAE related to AZD1775. | 0 | 8 | 9 | 7 | 1 | 1
  Pts. with ≥ one serious TEAE related to Chemo. | 0 | 8 | 9 | 7 | 1 | 1

13. Secondary Outcome: Serious Adverse Events Leading to Death
Description: The number of patients experiencing at least one serious adverse event (SAE) leading to death.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants
  No. with STEAE related to AZD1775 leading to death | 0 | 1 | 0 | 0 | 0 | 0
  No. with STEAE related to chemo leading to death | 0 | 1 | 0 | 0 | 0 | 0

14. Secondary Outcome: Treatment-Related Adverse Events Related to Adavosertib Leading to Treatment Discontinuation
Description: The number of patients experiencing at least one treatment-related adverse event related to adavosertib leading to treatment discontinuation.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 0 | 6 | 5 | 1 | 0 | 0

15. Secondary Outcome: Treatment-Related Adverse Events Related to Adavosertib Leading to Dose Reduction
Description: The number of patients experiencing at least one treatment-related adverse event related to adavosertib leading to dose reduction.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 2 | 18 | 5 | 11 | 0 | 0

16. Secondary Outcome: Treatment-Related Adverse Events Related to Adavosertib Leading to Treatment Interruption
Description: The number of patients experiencing at least one treatment-related adverse event related to adavosertib leading to treatment interruption.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 8 | 30 | 10 | 11 | 0 | 1

17. Secondary Outcome: Treatment-Related Adverse Events Related to Chemotherapy Leading to Treatment Discontinuation
Description: The number of patients experiencing at least one treatment-related adverse event related to chemotherapy leading to treatment discontinuation.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 0 | 6 | 5 | 1 | 0 | 0

18. Secondary Outcome: Treatment-Related Adverse Events Related to Chemotherapy Leading to Dose Reduction
Description: The number of patients experiencing at least one treatment-related adverse event related to chemotherapy leading to dose reduction.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 6 | 19 | 8 | 11 | 0 | 0

19. Secondary Outcome: Treatment-Related Adverse Events Related to Chemotherapy Leading to Treatment Interruption
Description: The number of patients experiencing at least one treatment-related adverse event related to chemotherapy leading to treatment interruption.
Time Frame: Throughout the duration of the study (up to 19 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
Number analyzed (Participants) | 9 | 38 | 23 | 12 | 6 | 6
Participants | 8 | 28 | 12 | 9 | 0 | 1

20. Secondary Outcome: Single Dose Adavosertib Cmax
Description: Maximum plasma concentration of adavosertib after a single oral dose (Cycle 1 Day 1) in combination with IV infusion of commonly used chemotherapy agents, including gemcitabine, paclitaxel, and carboplatin.
Time Frame: Pre-dose, 0.5 hr, 1 hr, 2 hr, 4 hr, 6 hr, and 8 hr
Population: The PK Analysis Set included all dosed patients who had at least one measurable plasma concentration collected post-dose which was obtained without any protocol deviation, violation, or other event which may have significantly affected the pharmacokinetics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Arm A 800 mg/m² Gemcitabine: Adavosertib175 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of 28 day cycles.
  Gemcitabine 800 mg/m² IV on Days 1, 8, and 15 of 28 day cycles.
- Arm A 1000 mg/m² Gemcitabine: Adavosertib 175 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of 28 day cycles.
  Gemcitabine 1000 mg/m² IV on Days 1, 8, and 15 of 28 day cycles.
Arm/Group | Arm A 800 mg/m² Gemcitabine | Arm A 1000 mg/m² Gemcitabine | Arm B | Arm C
Number analyzed (Participants) | 3 | 4 | 7 | 6
nM | 477.4 (3.776) | 571.1 (29.79) | 533.8 (37.29) | 556.6 (56.39)

21. Secondary Outcome: Multiple Dose Adavosertib Cmax
Description: Maximum plasma concentration of adavosertib after a multiple oral doses (Cycle 1 Day 3) in combination with IV infusion of 40 mg/m² pegylated liposomal doxorubicin.
Time Frame: Pre-dose, 1 hr, 2 hr, 4 hr, 6 hr, and 8 hr
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Arm D 175 mg: Adavosertib 175 mg orally BID (5 doses over 3 days) on Days 1-3 of 28 day cycles.
  Pegylated liposomal doxorubicin 40 mg/m² IV on Day 1 of 28 day cycles.
- Arm D 225 mg: Adavosertib 225 mg orally BID (5 doses over 3 days) on Days 1-3 of 28 day cycles.
  Pegylated liposomal doxorubicin 40 mg/m² IV on Day 1 of 28 day cycles.
Arm/Group | Arm D 175 mg | Arm D 225 mg
Number analyzed (Participants) | 5 | 4
nM | 4135 (65.8) | 23530 (30.15)

22. Secondary Outcome: Single Dose Adavosertib Tmax
Description: The time to reach maximum plasma concentration of adavosertib after a single oral dose (Cycle 1 Day 1) in combination with IV infusion of commonly used chemotherapy agents, including gemcitabine, paclitaxel, and carboplatin.
Time Frame: Pre-dose, 0.5 hr, 1 hr, 2 hr, 4 hr, 6 hr, and 8 hr
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Arm A 800 mg/m² Gemcitabine | Arm A 1000 mg/m² Gemcitabine | Arm B | Arm C
Number analyzed (Participants) | 3 | 4 | 7 | 6
hours | 2.00 [1.90 to 2.08] | 2.02 [0.50 to 4.05] | 4.08 [1.97 to 8.00] | 3.15 [1.75 to 4.07]

23. Secondary Outcome: Multiple Dose Adavosertib Tmax
Description: The time to reach maximum plasma concentration of adavosertib after multiple oral doses (Cycle 1 Day 3) in combination with IV infusion of 40 mg/m² pegylated liposomal doxorubicin.
Time Frame: Pre-dose, 1 hr, 2 hr, 4 hr, 6 hr, and 8 hr
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Arm D 175 mg | Arm D 225 mg
Number analyzed (Participants) | 5 | 4
hours | 3.92 [1.67 to 4.00] | 2.88 [1.87 to 4.00]

ADVERSE EVENTS:
Time Frame: Throughout the study, approximately 19 months
Arm/Group | Arm A | Arm B | Arm C | Arm C2 | Arm D-175 mg | Arm D-225 mg
All-Cause Mortality (participants affected / at risk) | 5/9 | 12/38 | 9/23 | 2/12 | 3/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/9 | 17/38 | 12/23 | 8/12 | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 9/9 | 38/38 | 23/23 | 12/12 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=9) | Arm B (N=38) | Arm C (N=23) | Arm C2 (N=12) | Arm D-175 mg (N=6) | Arm D-225 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (3) | 3 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraspinal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular Device Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=9) | Arm B (N=38) | Arm C (N=23) | Arm C2 (N=12) | Arm D-175 mg (N=6) | Arm D-225 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 (12) | 24 (82) | 13 (45) | 9 (48) | 3 (4) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (14) | 12 (25) | 5 (14) | 11 (51) | 1 (1) | 2 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 9 (12) | 11 (33) | 11 (90) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 2 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 8 (12) | 8 (9) | 1 (4) | 1 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (7) | 4 (4) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 31 (67) | 16 (33) | 6 (11) | 1 (1) | 5 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (9) | 23 (49) | 19 (38) | 10 (12) | 4 (5) | 4 (7)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 2 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7) | 19 (41) | 13 (24) | 4 (9) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (5) | 23 (33) | 17 (30) | 8 (11) | 3 (6) | 5 (5)
Oedema, Peripheral (General disorders) | 0 (0) | 10 (10) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 8 (11) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 6 (9) | 2 (3) | 1 (1) | 1 (1) | 1 (2)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (3) | 4 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 3 (5) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 4 (16) | 13 (64) | 5 (17) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 2 (10) | 7 (12) | 5 (19) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 2 (10) | 11 (64) | 4 (17) | 0 (0) | 1 (1) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (3) | 7 (9) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 6 (12) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (18) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 2 (8) | 3 (4) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 8 (13) | 6 (8) | 2 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (7) | 4 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4) | 3 (4) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 8 (8) | 7 (9) | 1 (1) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 8 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 6 (6) | 2 (5) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (12) | 4 (4) | 4 (6) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT02272790/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT02272790/SAP_001.pdf